CLINICAL TRIAL: NCT03733821
Title: Sleep Modifications in Patients With Cocaine Use Disorders Treated With Transcranial Magnetic Stimulation (TMS)
Brief Title: Subjective Sleep Quality in CUD TMS-Treated
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Novella Fronda (Other)
Collaborators: Studio Gallimberti Bonci & Partners (Unknown)
Responsible Party: Sponsor
Other Study IDs: SL33P0NCUDTM2TR34T3D
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Cocaine Use Disorder; Sleep Disturbance
Keywords: rTMS
MeSH Terms: conditions — Parasomnias | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CUD patients on HF-rTMS treatment: Patients fulfilling the Diagnostic and Statistical Manual of Mental Disorders - 5 (DSM 5) criteria for Cocaine Use Disorder undergoing a High Frequency rTMS protocol stimulating over the left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Non-invasive brain stimulation tool

SUMMARY:
Sleep disruptions are prevalent complaints in cocaine use disorder (CUD) subjects, either during consumption or withdrawal. Repetitive transcranial magnetic stimulation (rTMS) seem to be a promissing strategy in the treatment of chronic cocaine users.

The aim of this study will be to assess the variation on self-perceived sleep quality and drug use variables in individuals with CUD undergoing a rTMS protocol over the left dorsolateral prefrontal cortex (DLPFC).

DETAILED DESCRIPTION:
Cocaine use disorder (CUD) is a chronic relapsing brain disorder characterized by a problematic pattern of cocaine consumption leading to a clinically significant impairment. A core element of this disease is the increased vulnerability to relapse during the first weeks of abstinence. Commonly withdrawal symptoms as sleep disturbances, negative affect or craving, may contributes critically to relapses. Especially, sleep disruptions are frequently referred by CUD individuals during either use or abstinence. Moreover, polysomnographic (PSG) data demonstrate a worsening sleep during the first weeks of abstinence in chronic cocaine users, with diminishing rapid eye movement sleep (REM) time, reduction of total sleep time, increasing sleep latency, and chronically decreased slow-wave sleep (SWS) time. Such sleep anomalies appear to be durable and relate to the severity of withdrawal symptoms and clinical outcomes in the treatment of CUD. However, causality between sleep disturbances and CUD has not been clearly established yet. Interestingly, sleep deprivation and addictive substances have comparable neurobiological effects on several neurotransmitter pathways, particularly in the dopaminergic system. Therefore, the implementation of strategies to rewire the altered brain circuits might induce clinically significant improvements of addictive symptoms and the regulation of sleep patterns in CUD patients.

Recently, transcranial magnetic stimulation (TMS), an innovative and safe brain stimulation procedure, which induce neural electrical activity through the application of magnetic pulses over the scalp and with enduring effects on mood, has been applied as a promising therapeutic approach in addictive disorders. In fact, clinical pilot studies on CUD are giving preliminary support to the potential role of rTMS in decreasing cocaine craving and use. PSG studies in healthy volunteers have shown rTMS-induced changes in sleep architecture that are opposites to those found in CUD subjects, as a prolongation of REM latency or a marked increase in slow-wave sleep. The promising therapeutic effect of TMS on insomnia, restless legs syndrome and on sleep disturbances associated to epilepsy, depression and post-traumatic stress disorder has also been suggested. Further, rTMS application over DLPFC have revealed positives outcomes in patients with chronic primary insomnia, by reducing sleep latency, increasing the total sleep time and REM latency.

These findings suggest that rTMS might impact brain circuitry, modulating relevant functions as sleep architecture and potentially affecting addictive related symptoms as craving or negative affect.

The hypothesis of the present study is that rTMS treatment intervention might have a beneficial effect on sleep disturbances reported by CUD patients during the abstinence/withdrawal period. The investigators hypothesized also the positive outcome on accompanied cocaine withdrawal symptoms (as craving or mood) of rTMS.

Hence, the aims of the present study are:

1. to verify whether rTMS of the left DLPFC in CUD patients produces modifications on the subjective sleep quality patterns and drug use variables.
2. to further strengthen the results of previous CUD-TMS research, the investigators will test whether rTMS of the left DLPFC in CUD patients is safe and reduces cocaine use.

Procedures:

Patients with CUD will be evaluated for sleep disturbances, craving, depression, anxiety and other clinical symptoms by completing the following scales: Pittsburgh Sleep Quality Index (PSQI), Cocaine Craving Questionnaire (CCQ), Beck Depression Inventory-II (BDI-II), Self-rating Anxiety Scale (SAS), Alcohol Use Disorders Identification Test (AUDIT) and Symptoms checklist 90 - Revised (SCL-90-R). Participants could be undergo a battery of cognitive tests such as Wisconsin Card Sorting Test (WCST), Stop Signal Task (SST), Iowa Gambling Task (IGT), Stroop task or Delay Discounting Task (DDT). The pattern of drug use will be also monitored by recording drug use variables. The measures will be assessed before the rTMS treatment (baseline), and after 5 (Day 5), 30 (Day 30), 60 (Day 60) and 90 (Day 90) days during the treatment.

ELIGIBILITY:
Inclusion Criteria:

- Current diagnosis of CUD according to DSM-5;

Exclusion Criteria:

* Pregnancy or breastfeeding;
* Current DSM-5 diagnosis for Schizophrenia Spectrum and Other Psychotic Disorders, Major Depressive Disorder or Bipolar and Related Disorders;
* Current DSM-5 diagnosis for Alcohol and Substance use disorders (except Tobacco use disorders);
* Current DSM-5 diagnosis for Personality disorders;
* Current DSM-5 diagnosis for Primary Sleep-Wake Disorders;
* Prior history of un unstable medical illness, substantial neurological illness, any contraindication for rTMS (including implanted metal and devices in the body, and history of epilepsy);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants recruited after referral to specialty outpatient clinic Center for Addiction and meeting diagnostic criteria for Cocaine Use Disorder according to the Diagnostic and Statistical Manual of Mental Disorders - 5 (DSM 5), as assessed by an SUDs expert clinical psychiatrist.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
High frequency rTMS effects on subjective sleep quality in CUD patients | Baseline- Day 5 (after 10 rTMS sessions)- Day 30 (after 16 rTMS sessions)- Day 60 (after 24 rTMS sessions)- Day 90 (after 32 rTMS sessions)
  The subjective sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI). This scale is composed by 19 items clustered into 7 components, including sleep duration, sleep disturbance, sleep latency, daytime dysfunction, sleep efficiency, overall sleep quality, and sleep medication use. Each of them generates a score ranging from 0 to 3, with the highest value indicating the greatest dysfunction. The sleep component scores are summed to produce a global score ranging from 0 to 21 with the higher score indicating worse sleep quality. A global score higher than 5 is considered an indicator of relevant sleep disturbances.

SECONDARY OUTCOMES:
High frequency rTMS effects on self-reported craving in CUD patients | Baseline- Day 5 (after 10 rTMS sessions)- Day 30 (after 16 rTMS sessions)- Day 60 (after 24 rTMS sessions)- Day 90 (after 32 rTMS sessions)
  Self-reported craving will be assessed by Cocaine Craving Questionnaire (CCQ) which is a 5-item self-report questionnaire measuring five aspects of craving: current intensity, intensity during the previous 24 h, frequency, responsiveness to drug-related conditioned stimuli, and imagined likelihood of use if in a setting with access to drugs. Each craving aspects yields a score ranging from 0 to 9 with the highest values indicating high craving. The overall score is obtained by summing every item score and dividing it by 5. A higher mean craving score is associated with less likeliness to initiate abstinence.
High frequency rTMS effects on Depression Symptoms in CUD patients | Baseline- Day 30 (after 16 rTMS sessions)- Day 60 (after 24 rTMS sessions)- Day 90 (after 32 rTMS sessions)
  Depression symptoms will be assessed by Beck Depression Inventory - II (BDI - II) which is a 21-question multiple-choice self-report inventory with four options under each item, ranging from not present (0) to severe (3), measuring depressive symptoms. This inventory scoring is obtained by summing the highest ratings for each of the 21 items, with a sum scores range from 0 to 63. The severity levels suggested in the manual are the following: Scores between 0 and 13 indicate minimal, between 14 and 19 mild, between 20 and 28 moderate, and between 29 and 63 severe depression.
High frequency rTMS effects on Anxiety Symptoms in CUD patients | Baseline- Day 5 (after 10 rTMS sessions)- Day 30 (after 16 rTMS sessions)- Day 60 (after 24 rTMS sessions)- Day 90 (after 32 rTMS sessions)
  Anxiety symptoms will be assessed by Self-rating Anxiety Scale (SAS) which is is a 20-item measure developed to assess the frequency of anxiety symptoms based on diagnostic conceptualizations. It consists primarily of somatic symptoms. Each symptom is rated on a 4-point Likert scale on frecuency basis from 1 ('"none or a little of the time'") to 4 ('"most or all of the time''). Items 5, 9, 13, 17, and 19 are reversed scored and total scores on the SAS range from 0 to 80, with higher scores indicating more frequents anxiety symptoms.
High frequency rTMS effects on subjective symptoms of mental disorder in CUD patients | Baseline- Day 5 (after 10 rTMS sessions)- Day 30 (after 16 rTMS sessions)- Day 60 (after 24 rTMS sessions)- Day 90 (after 32 rTMS sessions)
  Subjective symptoms of mental disorder will be assessed by Symptoms checklist 90 - Revised (SCL-90-R) which is is a 90-item self-report inventory which assesses psychological distress in terms of nine primary symptom dimensions and three summary scores termed global scores. Each item describes a physical or psychological symptomthat is rated on a five-point scale ranging from 1 (not at all) to 5 (extremely). The Global Severity Index (GSI) is the single best indicator of the current level or depth of an individual's disorder. It combines information concerning the number of symptoms reported with the intensity of perceived distress.
High frequency rTMS effects on cocaine intake | Baseline- Day 5 (after 10 rTMS sessions)- Day 30 (after 16 rTMS sessions)- Day 60 (after 24 rTMS sessions)- Day 90 (after 32 rTMS sessions)
  Cocaine intake will be determined determined either via a urine drug test or referral reported relapse

CONTACTS AND LOCATIONS:
Overall Officials: Michela Sarlo, Assoc. Prof., Principal Investigator — Department of General Psychology, University of Padova; Nicola Cellini, PhD, Study Chair — Department of General Psychology, University of Padova; Stefano Cardullo, PhD, Study Chair — Fondazione Novella Fronda
Locations (1):
- Studio Gallimberti Bonci & Partners, Padua, Italy

REFERENCES:
- [Derived] Gomez Perez LJ, Cardullo S, Cellini N, Sarlo M, Monteanni T, Bonci A, Terraneo A, Gallimberti L, Madeo G. Sleep quality improves during treatment with repetitive transcranial magnetic stimulation (rTMS) in patients with cocaine use disorder: a retrospective observational study. BMC Psychiatry. 2020 Apr 6;20(1):153. doi: 10.1186/s12888-020-02568-2. PMID 32252720